## **Participant Informed Consent for Clinical Research**

**Study title for participants:** Study of Cemiplimab Combined with Dabrafenib and Trametinib in People with Anaplastic Thyroid Cancer

Official study title for internet search on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>: A Pilot Study of the Addition of Cemiplimab, an Antibody to PD-1, to the Treatment of Subjects with BRAF-Mutant Anaplastic Thyroid Cancer Who Are No Longer Responding to Dabrafenib and Trametinib

**Subtitle:** Group 2 (Dabrafenib/Trametinib at External Site)

Lead Researcher: Eric Sherman, MD (646-888-4234)

If you are the parent or legal guardian of the person who is being asked to participate in this research study, you may give consent on his or her behalf. The word "you" in this document refers to your child, if the participant is a minor, or to a person with a cognitive impairment for whom you are the Legally Authorized Representative (LAR).

## **Overview and Key Information**

### Why is this study being done?

We are asking you to take part in a clinical research study. We do research studies to try to answer questions about how to prevent, diagnose, and treat diseases like cancer.

You have anaplastic thyroid cancer, and you are receiving standard therapy with dabrafenib and trametinib.

This study is being done to see if adding the study drug, cemiplimab, to the standard therapy with dabrafenib and trametinib is an effective treatment against anaplastic thyroid cancer.

## Taking part in this study is your choice.

You can choose to take part or not to take part in this study, and you can change your mind at any time. Whatever choice you make, you will not lose access to your medical care or give up any legal rights or benefits.

This document presents important information to help you make your choice. Please take time to read it carefully. Talk with your doctor, family, or friends about the risks and benefits of taking part in this study. It's important that you have as much information as you need, and that all your questions are answered. See the *Where can I get more information?* section of this document for more information about research studies and for general information about cancer.

## What is the usual approach to my anaplastic thyroid cancer?

People who are not in a study are usually treated with more chemotherapy, or with a combination of dabrafenib and trametinib without cemiplimab. No treatments have been proven to be effective against anaplastic thyroid cancer after that cancer stops responding to dabrafenib and trametinib.



Approval date: 09-Nov-2021

## What are my other choices if I decide not to take part in this study?

- You may choose to have the usual approach described above
- You may choose to take part in a different research study, if one is available
- You may choose not to be treated for cancer
- You may choose not to be treated for cancer, but to receive comfort care to help relieve your symptoms

## What will happen if I decide to take part in this study?

If you decide to take part in this study, you will receive cemiplimab after your cancer does not appear to be responding to dabrafenib and trametinib alone. You will receive cemiplimab in addition to dabrafenib and trametinib, and you will receive the drug combination until your disease gets worse (progresses), or the side effects become too severe.

After you finish your study treatment, the study doctor and study team will watch you for side effects and follow your condition. You will come to the clinic for a physical exam and routine blood tests within 2 to 6 weeks of stopping treatment. After that visit, the study doctor and study team will call you or review your medical records every 3 months for 1 year.

## What are the risks and benefits of taking part in this study?

There are both risks and benefits to taking part in this study. It is important to think carefully about these as you make your decision.

#### Risks

We want to make sure that you know about a few key risks right now. We will also give you more information in the What risks can I expect from taking part in this study? section of this consent form.

If you choose to take part in this study, there is a risk that the study treatment may not be as good as the usual approach for your cancer at shrinking or stabilizing your cancer.

There is also a risk that you could have side effects from the study treatment. These side effects may be worse, and they may be different than you would have with the usual approach for your cancer.

Some of the most common side effects that the study doctors know about are:

- Fever
- Tiredness (fatigue)
- Nausea
- Vomiting
- Diarrhea

There may be some risks that the study doctors do not yet know about.

#### Benefits

Standard treatment with dabrafenib and trametinib has been shown to shrink or stabilize anaplastic thyroid cancer. It is not possible to know now if adding cemiplimab to the standard treatment will improve your response to treatment. Adding cemiplimab may help your cancer, or your cancer may stay



the same, or even get worse. However, what we learn from this research may help other people in the future.

## If I decide to take part in this study, can I stop later?

Yes, you can decide to stop participating in the study at any time.

The study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

If you decide to stop, let the study doctor know as soon as possible. It's important that you stop safely. This may mean slowly stopping the study treatment to avoid a sudden unsafe change or risk to your health.

If you stop, you can decide whether to let the study doctor or a member of the study team continue to contact you to ask questions about your health. We will not be able to withdraw information about you that has been used or shared with others before you informed us of your decision to stop.

## Are there other reasons why I might stop being in the study?

Yes. The study doctor may take you off the study if:

- Your health changes, and the study is no longer in your best interest
- New information becomes available, and the study is no longer in your best interest
- You do not follow the study rules
- For women who are able to have children: You become pregnant while you are in the study
- The study is stopped by the National Cancer Institute (NCI), Institutional Review Board (IRB), Food and Drug Administration (FDA), or the study sponsor, Memorial Sloan Kettering Cancer Center (MSK). The study sponsor is the organization that oversees the study.

It is important that you understand the information in this informed consent document before you make a decision about participating in this clinical trial. Please read, or have someone read to you, the rest of this document. If there is anything that you don't understand, ask the study doctor or nurse for more information.

## What is the purpose of this study?

This study will test whether adding the study drug, cemiplimab, to the standard therapy with dabrafenib and trametinib is an effective treatment against anaplastic thyroid cancer. The study will also look at how safe the drug combination is in participants.

When dabrafenib and trametinib are given to people whose cancers have mutations (changes) in the BRAF gene, the drugs prevent proteins made by the altered genes from sending signals to cancer cells. Without the signals, cancer cells stop growing and spreading. Participants in this study will have a mutation in the BRAF gene. Dabrafenib and trametinib have been used to treat other cancers in other research studies, and the FDA has approved this combination to treat anaplastic thyroid cancer.

Cemiplimab is a type of drug called a monoclonal antibody. Antibodies are made by the immune system to stick to and attack specific targets on cells. Cemiplimab blocks the protein PD-1 (programmed cell death receptor-1), which usually acts as a "brake" on the immune system. Blocking this protein is like releasing the brake, so the immune system can target cancer cells and destroy them. The FDA has



approved cemiplimab to treat certain types of skin cancer, but the FDA has not approved the drug for the treatment of your condition. Giving cemiplimab to people with anaplastic thyroid cancer is an investigational use of the drug. In addition, giving the combination of cemiplimab, dabrafenib, and trametinib to people with anaplastic thyroid cancer is an investigational use of the drugs.

The cemiplimab will be provided by Regeneron Pharmaceuticals, Inc.

About 15 people will take part in this study at Memorial Sloan Kettering Cancer Center (MSK).

### What are the study groups?

This study has two study groups. Participants in Group 1 will receive dabrafenib and trametinib first, and, if their cancer worsens, they will be treated with cemiplimab in addition to the standard treatment. Participants in Group 2 are already receiving dabrafenib and trametinib. Group 2 participants will receive cemiplimab, dabrafenib, and trametinib after their cancer does not appear to be responding to dabrafenib and trametinib alone.

This consent document is for Group 2 participants.

## What extra tests and procedures will I have if I take part in this study?

#### Before you begin the main part of the study:

The study doctor will review your medical records and the results of your exams, tests, and procedures to see if it is safe for you to take part in the study. This first part of the study is called screening. Most of the screening exams, tests, and procedures are part of the usual care that you would have if you were not in a study.

The tests and procedures that will be done only for research purposes, or that may be done more often because you are participating in this study, are listed below.

- Blood collection (about 2 teaspoons) for cell-free DNA (cfDNA) research testing, which will show
  whether altered (mutated) cancer genes in your tumor can also be found in your blood. Small
  pieces of genes free-floating in blood are called cell-free DNA (cfDNA). We will track the amount
  of cfDNA from your tumor that is found in your blood at different times before, during, and after
  treatment in this study. The amount of cfDNA may be related to your response to the treatment.
  This blood collection will occur at the same time as standard blood draws if possible.
- If you have stored (archival) tumor tissue available from a previous biopsy or surgical procedure at MSK or at an outside hospital, we will collect a piece of this sample for research testing.
- If your disease has not gotten worse while receiving dabrafenib and trametinib, you will have a tumor biopsy procedure to collect a small sample of your tissue for research testing. The sample will be used to study any genetic changes in your tumor, and why certain people respond to treatment while others do not. If you have stored (archival) tumor tissue available from a previous biopsy or surgical procedure, a piece of this sample may be collected instead.
  - You will sign a separate consent form for the biopsy procedure. The doctor doing the biopsy will explain what will happen, including any risks or possible side effects that may result from collecting the sample. More information about the risks of this procedure is provided in the What risks can I expect from taking part in this study? section of this consent form.
  - We will study your samples to improve our understanding of the way changes in genes can affect the risk of cancer and other diseases. Genes are the "blueprints" for our bodies.



Sometimes genes may have changes that occur during your lifetime that can affect the way a gene works. These changes (mutations) may cause cells to grow rapidly and abnormally, and become a cancer that you cannot pass on to your family members (somatic mutation). However, some people develop cancer because they were born with a mutation in a gene. People who develop cancer because of a genetic mutation usually inherit this genetic change from their mother or their father (germline mutation). Other family members (brothers, sisters, and children) may share this same mutation. Most people with cancer did not develop their disease because of an inherited mutation.

- We will look for changes in your genes using a test called Whole Genome Sequencing or Whole Exome Sequencing (WGS/WES). Your data may be used to learn more about cancer and other diseases. Data from large numbers of people can help researchers learn how changes in the order (sequence) of genes might affect a disease or a person's response to treatment, identify possible links between diseases, and provide new ideas for drug development and personalized therapies.
- After your research test samples have been studied, if any part of them is left over, the
  material will be stored for an indefinite period of time for use in future research. Your
  sample(s), including your DNA, may be used or stored for as long as they are useful for
  research purposes
- Neither you nor your doctor will be given the results of any genetic research testing done on your samples. If you or your family are interested in learning more about inherited risk factors for cancer, ask your study doctor for a referral to MSK's Clinical Genetics Service

#### During the study:

Each 21-day treatment period is called a Cycle. You will take the following drugs at home, by mouth:

- Dabrafenib capsules twice a day, at least 1 hour before or 2 hours after a meal
- Trametinib tablets once a day, at least 1 hour before or 2 hours after a meal

A member of the study team will give you a pill diary, so that you can write down, every day, when you take dabrafenib and trametinib. Instructions about how to take the study treatment are included in the pill diary. Bring your completed diary to all your study appointments, and bring your medication bottle(s), even if the bottle is empty

You will receive the study drug, cemiplimab, as an intravenous infusion through a needle placed in a vein in your arm on Day 1 of each Cycle. The cemiplimab infusion will take about 30 minutes.

You will receive cemiplimab, dabrafenib, and trametinib until your disease gets worse (progresses), or the side effects become too severe.

If some or all of your tumors are progressing and they can be treated with radiation therapy, and the study doctor believes you are benefiting from the study treatment, you may be able to stay in the study while you are receiving radiation therapy, as long as the therapy does not take more than 4 weeks.

If you require radiation therapy during this study, you will not take dabrafenib or trametinib from 1 week before starting radiation therapy until 1 week after you complete the therapy.

Exams, Tests, and/or Procedures



You will have tests and procedures during the main study. The procedures that will be done only for research purposes, or that may be done more often because you are participating in this study, are listed below.

- Blood Collection (about 2 teaspoons) for plasma-free DNA research testing. This blood collection will occur at the same time as standard blood draws if possible.
- Tumor biopsy procedure, to collect a small sample of your tissue for research testing, within 4
  weeks of starting cemiplimab treatment, and 2 to 6 weeks after starting cemiplimab
  - You will sign a separate consent form for the biopsy procedure. The doctor doing the biopsy will explain what will happen, including any risks or possible side effects that may result from collecting the sample.
  - o If you are scheduled for a surgery or biopsy that will be done as standard of care while receiving treatment on the study, tissue may be collected for research testing. This will either be in addition to the above mentioned timepoints, or to take the place of one of the above mentioned timepoints. Your treating doctor will discuss the collection process with you.

#### **End-of-Treatment and follow-up visits:**

You will come back to the clinic for a physical exam and routine blood tests within 2 to 6 weeks of your last treatment for the End-of-Treatment visit. After this visit, you will not need to return to the clinic. The study doctor or study team will call you or review your medical records every 3 months for 1 year to check on your health.

A Study Calendar that shows how often you will have these exams, tests, and procedures is provided at the end of this consent form. The calendar also includes exams, tests, and procedures that are part of your usual care.

#### Will I receive the results of my research tests?

Neither you nor your doctor will receive the results of any tests done for research purposes during this study.

## What risks can I expect from taking part in this study?

If you choose to take part in this study, there is a risk that:

- You may lose time at work, school, or at home, and you may spend more time than usual in the hospital or doctor's office
- You may be asked sensitive or private questions that you do not usually discuss
- There may be a risk in finding out new genetic information about yourself. New health information about inherited traits that might affect you or your family (blood relatives) could be found during a research study.

The drugs used in this study may affect how different parts of your body work, such as your liver, kidneys, heart, and blood. The study doctor will be testing your blood throughout the study, and he or she will let you know if changes occur that may affect your health.

There is also a risk that you could have side effects from the study treatment/study approach.

Important information about side effects:

The study doctors do not know who will or will not have side effects.



- Some side effects may go away soon, some may last a long time, and some may never go away.
- Some side effects may make it difficult for you to have children.
- Some side effects may be mild. Others may be very serious, and may even result in death.

Important information about how you and the study doctor can make side effects less of a problem for you:

- If you notice or feel anything different, tell the study doctor. He or she can check to see if you are having a side effect.
- The study doctor may be able to treat some side effects.
- The study doctor may adjust the study drugs to try to reduce your side effects.

The tables below show the most common and the most serious side effects that researchers know about. There may be other side effects that the doctors do not yet know about. If important new side effects are found during this study, the study doctor will discuss them with you.

#### Possible side effects of dabrafenib and trametinib:

#### Common, some may be serious

In 100 people receiving dabrafenib and trametinib, more than 10 and as many as 100 may have:

- Fever, which may be associated with low blood pressure, dehydration, dizziness, and/or fainting
- Bleeding (hemorrhage), or major bleeding events, defined as symptomatic bleeding in a critical area or organ including the brain. A bleeding event may require you to be admitted to the hospital and receive surgery.
- Chills
- Decreased appetite
- Headache
- Dizziness
- Cough
- Stomach area (abdominal) pain
- Constipation
- Diarrhea
- Nausea
- Vomiting
- Skin effects, which may include rash, dryness, and/or itching
- Pain or stiffness of joint(s)
- Muscle pain
- Pain in arms or legs
- Feeling weak or tired
- Swelling of your arms and/or legs (peripheral edema)
- Abnormal liver tests (ALT increased, AST increased), which may mean that your liver
  is not working normally. This condition is usually mild and reversible, but it may be
  serious or life-threatening. Your study doctor will check your liver tests regularly while
  you are receiving the study treatment. Tell your study doctor or study nurse if you have



#### Common, some may be serious

In 100 people receiving dabrafenib and trametinib, more than 10 and as many as 100 may have:

itching, yellowing of the eyes or skin, dark urine, or pain or discomfort in the right upper area of your stomach.

- High blood pressure
- Inflammation of the throat and nasal passage (nasopharyngitis)

#### Occasional, some may be serious

In 100 people receiving dabrafenib and trametinib, between 1 and 10 may have:

- A type of skin cancer called squamous cell carcinoma (SCC)
- Thickening of the skin on the palms of your hands and soles of your feet, which may also be tender or painful, with a burning feeling (hand-foot skin reaction)
- Skin effects, which may include thickening of the skin (hyperkeratosis), skin cracking, warts (papilloma), wart-like growths (seborrhoeic keratosis), skin lesions, acne-like rash, scaly patches (actinic keratosis), redness, rash with pus-filled lesions, and/or inflammation of the fatty layer under the skin, which can cause red, painful lumps (panniculitis)
- Skin infection (cellulitis)
- Dry mouth
- Dehydration
- Night sweats
- Muscle spasms
- Bladder infection
- Nail problems, including pain, infection, and swelling of the cuticles (paronychia)
- Low number of platelets, which may cause bleeding and bruising (thrombocytopenia)
- A decrease in red blood cells, which may cause tiredness, shortness of breath, or dizziness (anemia)
- Low blood sodium (salt) level, often associated with dehydration (hyponatremia)
- Low phosphate level, which may cause muscle weakness (hypophosphatemia)
- High blood sugar (hyperglycemia) or excess sugar in the blood; if severe, this condition may require you to be admitted to the hospital and receive urgent treatment (diabetes)
- Decrease in the number of white blood cells, which may lead to increased risk of infection and can be life-threatening (leukopenia)
- Low blood pressure, which may cause dizziness, lightheadedness, or fainting
- Facial swelling
- Shortness of breath (dyspnea)
- Redness, swelling, or pain in the mouth (stomatitis)
- Hair loss
- Kidney failure: Your blood pressure rises and harmful wastes build up in your body.
   You may have tiredness (fatigue), nausea, and loss of appetite. This condition can be serious or life-threatening. If you have kidney failure, you will need treatment, such as dialysis (removing waste products and excess fluid from the body), to make up for the loss of kidney function.



#### Occasional, some may be serious

In 100 people receiving dabrafenib and trametinib, between 1 and 10 may have:

- Swelling of and/or redness and/or pain in the lining of the mouth or nose, or sometimes around the eyes (mucosal inflammation)
- Flu-like illness
- Inflammation of one or more hair follicles (folliculitis)
- Increased blood level of protein (blood creatine phosphokinase increased)
- Decreased heart rate (bradycardia), which can cause dizziness, fainting, and tiredness
- Changes in how well the heart pumps blood (decreased ejection fraction), which may cause an irregular heartbeat, heart failure, shortness of breath, swelling in your legs, or tiredness

#### Rare, and serious

In 100 people receiving dabrafenib and trametinib, 1 or fewer may have:

- Allergic reaction
- New melanomas
- Skin tags or noncancerous (benign) skin growths that some people develop as they age (acrochordon)
- Problems with your eyes, including inflammation of the eye (uveitis), swelling around the eyes (periorbital edema), or separation of the light-sensitive layer of the eye (the retina) from its supporting layers (retinal detachment, chorioretinopathy), which can result in blurry vision. These vision problems often improve; however, there is a slight risk that they may not improve and could lead to blindness.
- The heart is not able to pump blood properly, or it has difficulty filling with blood (cardiac failure, left ventricular dysfunction), which can cause weakness and tiredness, swelling, and shortness of breath.
- Inflammation of the pancreas, a gland that controls blood sugar levels and helps digest food. This condition could cause pain in the upper abdomen, and may become severe, causing nausea and vomiting, fever, and rapid heart rate. This could require you to be admitted to the hospital and may be life-threatening.
- Breakdown of muscle, which can lead to muscle pain and kidney damage (rhabdomyolysis)
- Inflammation of the lung tissue (pneumonitis or interstitial lung disease) may cause shortness of breath and changes in chest CT scans

## Possible side effects of cemiplimab:

#### Common, some may be serious

In 100 people receiving cemiplimab, more than 10 and as many as 100 may have:

- Fatigue
- Rash
- Diarrhea



#### Occasional, some may be serious

In 100 people receiving cemiplimab, between 1 and 10 may have:

- Nausea
- Vomiting
- Constipation
- Abdominal pain
- Dry mouth
- Inflammation of mouth and lips (stomatitis)
- Difficulty swallowing (dysphagia)
- Fever
- Chills
- Flu-like illness
- Swelling of an arm or leg
- Cough
- Shortness of breath
- Inflammation of the lung (pneumonitis)
- Joint pain (arthralgia)
- Muscle pain (myalgia)
- Decreased appetite
- Decreased weight
- Dehydration
- Itching
- Low phosphate in the blood (which does not cause symptoms but causes an abnormal blood test)
- Low red blood cells that can cause tiredness (anemia)
- Low white blood cells (which can make it more likely for you to get an infection)
- Damage to the liver (from inflammation) that does not cause symptoms but causes an abnormal result on a blood test of liver function
- Headache
- Underactive or overactive thyroid gland (which can cause tiredness, constipation, hair loss, sensitivity to heat or cold temperatures, mood changes, sweating, muscle aches, a fast heartbeat, or weight changes)
- Diabetes
- Infusion reaction (similar to an allergic reaction) that occurs during or shortly after the infusion; symptoms include fever and chills, skin rash or swelling at the infusion site, nausea, vomiting, headache, cold-like symptoms, difficulty breathing, and low blood pressure
- Trouble sleeping (insomnia)

#### Rare, and serious

In 100 people receiving cemiplimab, 1 or fewer may have:

• Encephalomyelitis (inflammation of the brain), which may result in severe memory loss and occasionally death



#### Rare, and serious

In 100 people receiving cemiplimab, 1 or fewer may have:

- Myasthenia gravis, a disease that causes muscle weakness
- Inflammation of the colon (colitis), which may cause diarrhea, abdominal pain, rectal pain, rectal bleeding, weight loss, or fatigue
- A narrowing of air passages in the lungs, causing shortness of breath (bronchospasm)
- Diabetic ketoacidosis, a severe complication of diabetes (high blood sugar) where the body makes too much acid in the blood
- Toxic epidermal necrolysis (Lyell's syndrome), a life-threatening reaction to a medicine. Lyell's syndrome can cause painful blisters or red or purple discoloration anywhere on your skin (which may look like a burn and may peel off); swelling in the face or tongue; or watery, red, and burning eyes.

**Possible risks and discomfort associated with research biopsies**: Risks associated with biopsies include pain, redness, swelling, bleeding, bruising, infection, and, rarely, death. The doctor performing the biopsy will explain the details and risks of the procedure, which may vary, depending on how the biopsy sample will be obtained. You will sign a separate consent document before you undergo this procedure.

**Possible risks of radiation-based diagnostic imaging:** You will be exposed to low amounts of radiation from the imaging procedures performed during this research study. The imaging procedures involve using a CT scan to guide the biopsy procedure. The radiation exposure from these procedures is considerably lower than the exposure associated with other standard-of-care imaging procedures. Each year, many thousands of patients routinely undergo similar procedures and receive similar doses of radiation with no short- or long-term adverse effects.

**Possible risks of contrast materials:** Contrast materials, also called contrast agents or contrast media, are injected into a vein in the arm to improve the pictures produced by CT scans. Contrast materials are generally very safe, but adverse reactions ranging from mild to severe may occur. Serious allergic reactions or other reactions are rare. A small percentage of patients may develop a delayed allergic reaction, with a rash that can occur hours to days after the injection of the contrast agent. Most of these rashes are mild, but severe rashes may require medication; please discuss any reactions with the study doctor.

**Reproductive risks**: You should not get pregnant, breastfeed, father a baby, or donate sperm while you are in this study. The drugs used in this study could be very damaging to an unborn baby. Check with the study doctor about what types of birth control or pregnancy prevention to use while you are in this study. Male participants must continue to use these methods for 6 months after their last dose of cemiplimab.

Let the study doctor know about any questions you may have about possible side effects. You can ask the study doctor questions about side effects at any time.

## What are my responsibilities in this study?

If you choose to take part in this study, you will need to:

Keep your study appointments



- Tell the study doctor about:
  - o All medications and any supplements you are taking
  - Any side effects from these medications or supplements
  - Any doctor visits or hospital stays outside of this study
  - Whether you have been or are currently in another research study
- Remember to bring your completed pill diary to all your clinic appointments, along with your medication bottle(s), even if the bottle is empty.
- Avoid products made with grapefruit, grapefruit juice, Seville oranges, pomelos, exotic citrus fruits, or grapefruit hybrids during the study. These products may affect the way dabrafenib works.

## Is there a conflict of interest for this study?

This study is sponsored by Memorial Sloan Kettering Cancer Center and funded by Regeneron Pharmaceuticals, Inc. One of the investigators involved in this study has an ownership interest (such as stock or stock options) in Regeneron. The amount of this financial interest might be affected by the results of the study. This means that the investigator could gain or lose money, depending on the results of the study. If you would like to know more about the steps MSK has taken to protect your best interests while you are in this study, please contact the MSK Patient Representative Department at 212-639-7202.

## What are the costs of taking part in this study?

You will not have to pay for the cemiplimab or for tests and procedures done only for research purposes, including:

- Tumor biopsy procedures (all times you have biopsies) unless the tissue is being obtained due to standard of care
- Plasma-free DNA research testing using blood collected at the screening visit, during study treatment, and at the End-of-Treatment Visit

It is possible that cemiplimab may not continue to be supplied while you are in the study. This possibility is unlikely, but if it occurs, your study doctor will talk with you about your options.

You and/or your health plan/insurance company will have to pay for all the other costs of treating your cancer while you are in this study. These charges include the costs of dabrafenib and trametinib, insurance co-pays and deductibles, as well as tests, procedures, or drugs that you get during the study to monitor your safety, and to prevent or manage any side effects.

Although you do not have to pay for the study drug, the cost of getting the cemiplimab ready and giving it to you is not paid by the study sponsor, so you or your insurance company may have to pay for this.

Talk to your insurance provider and make sure that you understand what your insurance pays for and what it does not pay for if you take part in this clinical trial. Also find out if you need approval from your health plan before you can take part in this study.

The study doctor or nurse can help you find the right person to talk to if you are not sure which costs will be billed to you or your insurance provider.



## Will I receive payment for taking part in this study?

You will not be paid for taking part in this study.

Your biospecimens (blood, tissue) may be used in the development of new tests, drugs, or other products for sale. If they are, you will not receive any payment from the sale of these products.

## What happens if I am injured or hurt because I took part in this study?

You will get medical treatment if you are injured as a result of taking part in this study.

If you think that you have been injured as a result of taking part in this research study, tell the study doctor or the person in charge of the study as soon as possible. The name and telephone number of the person in charge of this research are listed on the first page of this consent form.

We will offer you treatment for research injuries that happen as a result of your taking part in this study. You and/or your health plan will be charged for this treatment. Medical services will be offered at the usual charge. You will be responsible for any costs not covered by your health plan/insurance company.

If you think that your injury was a result of medical error, you keep all your legal rights to receive payment for treating the injury, even though you are in a study.

### Who will see my medical information?

Your privacy is very important to us, and the researchers will make every effort to protect it. Trained staff at Memorial Hospital may review your records, if necessary.

Access to your protected health information will be limited to those listed in the Research Authorization form, which is a part of the informed consent process.

Your information may be given out, if required by law. For example, some states require doctors to make a report to the state health board if they find that a participant in a research study has a contagious disease like tuberculosis. However, the researchers will do their best to make sure that any information about you that may be released will not identify you.

In the future, your information (data) and biospecimens may be de-identified, which means that your data and/or biospecimens will be assigned a unique code, and the list that links the code to your name will be stored separately from your biospecimens and data. Your de-identified information and biospecimens may be used for research that has not been described in this consent form, and they may be shared with another investigator for future research. You will not be asked if you agree to take part in future research studies.

If your information from this study is used in any reports or publications, your name and anything else that could identify you will not be used. It is possible that your de-identified information from this study will be shared with other researchers outside of MSK. All requests for data sharing will be reviewed by MSK, and if individual results are included in the data, they will not contain any identifiable information about you, such as your name, address, telephone number, or social security number. Your privacy is very important to us and we use many safety procedures to protect your privacy. However, we cannot guarantee that no one will ever be able to use your information to identify you.



A Federal law, the Genetic Information Nondiscrimination Act (GINA), generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that we get from this
  research when making a decision to hire, promote, or fire you, or when setting the terms of your
  employment.

Be aware that this Federal law does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, long-term care insurance, or if you are a member of the military.

## Where can I get more information?

You may visit the NCI web site at <a href="http://cancer.gov/">http://cancer.gov/</a> for more information about research studies, or for general information about cancer. You may also call the NCI Cancer Information Service to get the same information at 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

You can talk to the study doctor about any questions or concerns that you may have about this study, or to report side effects or injuries. You may also contact the lead researcher listed on the first page of this consent.

For questions about your rights while you are participating in this study, call the MSK Institutional Review Board (IRB) at 212-639-7592. If you have concerns, complaints, or input on research, or if you would like more information about the informed consent process, please contact the MSK Patient Representative Department at 212-639-7202.



## Research Authorization for the Use and Disclosure of Protected Health Information (PHI)

Study of Cemiplimab Combined with Dabrafenib and Trametinib in People with Anaplastic Thyroid Cancer: Group 2

Federal law requires Memorial Sloan Kettering Cancer Center (MSK) to protect the privacy of information that identifies you and relates to your past, present, and future medical conditions (protected health information; PHI). We are committed to protecting the privacy of your information.

If you enroll in this research study, your protected health information will be used and shared with others, as explained below. MSK must obtain your permission before using or sharing your protected health information for research purposes. This form helps to make sure that you are informed of the ways in which your information will be used or shared in the future.

Carefully read the information below before you sign this form. By signing this form, you agree to the use and disclosure of your information for this research study.

## 1. What protected health information about me will be used or shared with others during this research?

- Your medical records
- Your research records, including new health information created from study-related tests, procedures, visits, and/or questionnaires
- Any health information or clinical data associated with your biospecimens, if the information or data could be reasonably used to identify you. This information or data will be shared only if you have agreed to it by signing this informed consent document.
- HIV-related information, including any information indicating that you have had an HIV-related test; or that you have HIV infection, HIV-related illness, or AIDS; or any information that could indicate that you may have been exposed to HIV. (New York State requires us to obtain your consent to use or share this information.)

## 2. Who will use or share my protected health information?

MSK will use and share your protected health information. People and offices that deal with research oversight, quality assurance, and/or billing will be able to use and share your protected health information, including:

- The study's Principal Investigator and Co-Principal Investigators: Eric Sherman, MD; David Pfister, MD; and Alan Ho, MD, PhD
- Your research team at MSK, including the participating investigators, research staff, research nurses, fellows/residents, and clerical support staff
- Any healthcare personnel who provide services to you in connection with this study
- Members and staff of MSK's Institutional Review Board (IRB) and Privacy Board (PB)
- Staff of MSK's Clinical Research Administration, which oversees clinical studies, and Clinical Research Information Technology Group, which manages research databases
- Members of MSK's Data Safety Monitoring Board/Committee and the Quality Assurance Committee



## 3. With whom outside of MSK may my protected health information be shared?

Although all reasonable efforts will be made to maintain the confidentiality of your protected health information, it may be shared with and used by the following:

- The company or organization that provides the drug (cemiplimab) for the study, Regeneron Pharmaceuticals, Inc.
- MSK's research collaborators, business partners, subcontractors and agent(s), in the United States or in other countries, working to conduct the study, to monitor the study, or to analyze the study information for this study or for other research about the study drug
- Other research doctors and medical centers participating in this research.
- Federal and state agencies, and other domestic or foreign government bodies, if required by law and/or necessary for oversight purposes, including:
  - Office for Human Research Protections (OHRP) of the US Department of Health and Human Services (HHS)
  - US Food and Drug Administration (FDA) and other regulatory agencies responsible for oversight of research
  - National Cancer Institute (NCI)/National Institutes of Health (NIH)
- Other qualified researchers, approved by Memorial Sloan Kettering Cancer Center, who may receive individual research results that do not identify you.

Some of the organizations that may receive your protected health information may not have to satisfy the privacy rules and requirements; they may share your information with others without your permission.

## 4. Why will my protected health information be used by or shared by MSK or others?

The main reasons for the use or sharing of your information include the following:

- To conduct the study, to monitor your health status, to measure the effects of the drug(s)/device(s)/procedure(s) being studied, and to determine the research results
- To ensure that the research meets legal and institutional requirements
- To develop new tests, procedures, and commercial products
- To enhance research databases, so that scientists can design better research studies to develop new therapies for patients and to gain a better understanding of disease
- To assist with MSK medical treatment, billing, or healthcare operations. For example, medical information produced by this research study will become part of your hospital medical record.

## 5. For how long will my protected health information be used or shared with others?

There is no set date at which your protected health information that is being used or shared for this research study will be destroyed or no longer used. The information used and created during the



study may be analyzed for many years, and it is not possible to know when this analysis will be completed.

## 6. Statement of privacy rights:

- It is your right to refuse to sign this authorization form. If you do not sign this form, you will not be able to participate in this research study. However, if you do not sign, it will not affect your ongoing medical treatment or healthcare coverage.
- You have the right to withdraw your permission for MSK to use or share your protected health information. Please note that we will not be able to withdraw all the information about you that already has been used or shared with others to carry out research-related activities such as oversight, or information that is needed to ensure the quality of the study. To withdraw your permission, write to the study doctor listed on the first page of this consent form at: Memorial Sloan Kettering Cancer Center, 1275 York Avenue, New York, NY 10065. If you withdraw permission for us to use or share your protected health information, you will not be able to continue to participate in this research study.
- You have the right to request access to your protected health information that is being used or shared during this research and that is related to the research or to payment for the research. However, you may access this information only after the study is completed. You may have access to your medical record at any time. To request this information, please contact the study doctor whose name and telephone number are listed on the first page of this consent form. You may also ask the study doctor to correct any study-related information about you that is wrong.

#### Notice concerning HIV-related information

Individuals/organizations are prohibited from sharing any HIV-related information about you without your approval, unless they are permitted to do so under federal or state law. You have a right to request the list of people who may receive or use your HIV-related information without your authorization.

If you experience discrimination because of the release or disclosure of your HIV-related information, you may contact the New York State Division of Human Rights at 888-392-3644 or the New York City Commission on Human Rights at 212-306-7500. These agencies are responsible for protecting your rights.



## Participant Informed Consent/Research Authorization for Clinical Research

### Statement of professional obtaining consent

I have fully explained this clinical research study to the participant or to his/her Legally Authorized Representative (LAR). In my judgment, and in that of the participant or his/her LAR, sufficient information, including risks and benefits, was provided for the participant or his/her LAR to make an informed decision. The consent discussion will be documented in the participant's EMR.

| The consent discussion will be | | · |
|---|---|---|
| Consent | ing profess | sional must personally sign and date |
| Consenting professiona | al's | Date: |
| signature | | |
| Consenting professiona (Print) | ıl's name | |
| I have read this form that desc<br>with the consenting profession<br>this clinical research study; (2)<br>information (data about myself<br>of this consent form. | ribes the clin<br>lal. By signing<br>to authorize<br>f/the participa | Representative's [LAR's)]) statement ical research study. I have also talked it over to my satisfaction g below, I agree to the following: (1) to voluntarily participate in the use and disclosure of my/the participant's protected health int); and (3) to state that I have received a signed and dated copy |
| | icipant/L/ | AR must personally sign and date |
| Participant/LAR | | Date: |
| signature Participant/LAR | | |
| name (Print) | | |
| LAR relationship to | | |
| participant | | |
| VAT' to a series of the series (if the | | |
| participant's (or LAR's) lan for the participant (or LAR) Other: I confirm that the co | peaking partic<br>guage, and I<br>onsent discus | cipant: I declare that I am fluent in both English and in the confirm that the consent discussion was appropriately interpreted assion occurred, and that the participant agreed to participate in his/her mark, or verbally agreeing. |
| Name of witness: | | |
| <b>Signature of witness:</b> (The name of the witness mus | | ented in the EMR.) |
| Interpreter (if required Name of interpreter (if | present):_ | |
| ID number (if phone int | | |
| (The interpreter's name or ID i | number must | be documented in the EMR.) |

The participant/Legally Authorized Representative must be provided with a signed copy of this form.



## Study Calendar:

This calendar shows the exams, tests, and procedures that will be done as part of this research study, as well as the tests and procedures that are part of your usual care.

| | | ı | | T | 1 | 1 | 1 |
|---|---|---|---|---|---|---|---|
| | Screening<br>(28 days) | Cycle 1<br>Day 1 | Cycle 2<br>Day 1 | Cycle 3 Day 1 & odd Cycles | Cycle 4 Day 1 & even Cycles | End-of-<br>Treatment<br>visit | Long-term<br>follow-up |
| Medical history | Х | | | | | | |
| Physical exam and vital signs | X | Х | Х | Х | Х | Х | |
| Routine blood tests | Х | Х | Х | X | Х | Х | |
| Pregnancy test, if applicable | Х | | | | | | |
| Electrocardiogram | Х | | | | | Х | |
| Echocardiogram or MUGA scan | Х | | | | | | |
| Eye exam | X | | | | | | |
| CT or MRI scans | Х | | | Х | | Х | |
| Collection of stored (archived) tissue | Х | | | | | | |
| Tumor biopsy procedure <sup>1</sup> | Х | | X | | | | |
| Research Blood Test | Х | X | | | | Х | |
| Trametinib (once daily) | | Х | Х | Х | Х | | |
| Dabrafenib (twice daily) | | Х | Х | Х | Х | | |
| Medication diary review for dabrafenib & trametinib | | Х | Х | X | × | х | |
| Cemiplimab infusion | | Х | Х | Х | Х | | |
| Review of medications and side effects | Х | | l | | | | |
| Phone call or review of medical records to check condition | | | | d of care biopey ma | | | Every 3<br>months<br>for 1 year |

<sup>1.</sup> A standard of care surgery or standard of care biopsy may be used for a given timepoint

